CLINICAL TRIAL: NCT06705283
Title: Effects Of Yoga And Whole Body Vibration Training On Women With Stress Urinary Incontinence
Brief Title: Yoga and Vibration Training for Stress Urinary Incontinence in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Pinar Yasar, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 78/30
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; yoga; whole body vibration training; pelvic floor muscle; quality of life
MeSH Terms: conditions — Urinary Incontinence | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- yoga group (Experimental): This is a group where yoga and home exercise (pelvic floor muscle training) will be done together.
  Interventions: Procedure: yoga and home exercise
- whole body vibration training (WBVT) group (Experimental): This is a group where whole body vibration training and home exercise (pelvic floor muscle training) will be done together.
  Interventions: Procedure: whole body vibration training and home exercise
- home exercise group (Active Comparator): This is a group where pelvic floor muscle training will be done.
  Interventions: Procedure: home exercise group

INTERVENTIONS:
Procedure: yoga and home exercise — The intervention period for the study was determined as 6 weeks. It has been decided that yoga practice will be done 3 times a week for 45 minutes.
  Poses to be practiced in the yoga group:
  1. Tadasana (mountain pose)
  2. Utkatasana (chair pose)
  3. Trikonasana (triangle pose)
  4. Malasana (squat pose):
  5. Viparita Karani Variation (legs up the wall pose)
  6. Salamba Set Bandhasana (supported bridge pose)
  7. Supta Baddha Konasana (reclining bound angle pose)
  8. Savasana (dead pose)
  Arms: yoga group
Procedure: whole body vibration training and home exercise — A total of 40-45 minutes of training was planned for WBVT, including warm-up (10 minutes), active phase (25-30 minutes) and cooling phase (5 minutes).
  Arms: whole body vibration training (WBVT) group
Procedure: home exercise group — Pelvic floor muscle training will be done in the home exercise group. This training will be done in the form of slow and fast contractions of the pelvic floor muscles in supine, chin up, sitting, squat and standing positions.
  Arms: home exercise group

SUMMARY:
This study aimed to compare the effects of yoga and Whole Body Vibration Training on pelvic floor muscle strength, severity of urinary symptoms and UI-related quality of life in women with UI.

The intervention period for the study was determined as 6 weeks. It has been decided that yoga practice will be done 3 times a week for 45 minutes, and whole body vibration training will be done for 45-55 minutes. The home exercise group will perform the planned exercise protocol every day for 6 weeks.

The results of the study will be evaluated by statistical analysis as a result of the interventions and evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-60,
* patients with SUI or Mix UI with a predominant SUI component,
* patients who have not received treatment with any physical therapy modality in the last 3 months,
* patients who signed the informed consent form.

Exclusion Criteria:

* Those with neurological diseases that may cause incontinence
* Those with prolapse
* Those using intrauterine devices
* Obesity (BMI >30)
* Patients with serious systemic diseases that prevent them from exercising (Cardiovascular disease, COPD, CVO and/or cancer)
* Patients with pure urge or mixed UI with a predominant urge component
* Patients with a history of thrombosis
* Patients who engage in high-intensity sports activities for at least half an hour at least twice a week (tennis, aerobic exercise, running, exercises with body weight).
* Patients with neurological or vestibular disease that may cause balance disorders
* Patients with grade 3 or 4 knee and/or hip osteoarthritis
* Patients with a history of knee and/or hip joint replacement surgery
* Patients with kidney or gallbladder stones
* Patients with acute disc herniation or spondylolisthesis

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
pelvic floor muscle strength test | 6 weeks
  Pelvic floor muscle strength evaluation will be performed with a perineal EMG biofeedback device with a vaginal probe. After the pressure probe is inserted into the vagina, the patient will be asked to contract the pelvic floor muscles. Contractions will be repeated 3 times and averaged. The obtained value will be recorded in cmH2O.
Numerical Rating Scale | 6 weeks
  It is used for severity of urinary incontinence. The participant was asked "How much urine do you think you leak?" The question will be asked and the student will be asked to make a mark on the chart that scores between 0-10 points.0 means no urine leakage, 10 means a lot of urine leakage.
International Consultation of Incontinence Society-Short Form | 6 weeks
  The scale addresses the frequency of UI and how much UI affects a person's life. There are a total of 4 questions, 3 of which are included in the scoring. A total of 0-21 points are given (0: no leakage, 1-5: mild, 6-12: moderate, 13-18: severe, 21: serious urine leakage). As the score increases, the severity of UI and the impact on quality of life increase.
1 hour pad test | 6 weeks
  • Pad test is an easy-to-perform test that determines the severity of urine leakage objectively. During the implementation of this test, the protocol established by the International Continence Society will be taken as basis. The steps of the protocol are as follows: 0. min: The weight of the clean pad is weighed. It is given to the patient. After wearing the pad, the patient is asked to drink 500 ml of water in a short time.
  30 min: walking and climbing stairs 45th minute: Coughing 10 times, sitting down and standing up 10 times, picking up something from the ground 10 times, jumping 10 times, washing hands under running water for 1 minute, running for 1 minute.
  60th minute: Weighing the pad taken from the patient again. After the evaluation steps are completed, the amount of urine leakage is calculated by subtracting the weight of the clean pad from the weight of the used pad.
Incontinence Impact Questionnaire-7 | 6 weeks
  There are 7 items in the scale. Items are scored between 0-3, resulting in a total score between 0-21. It is understood that as the score obtained from the scale increases, the severity of UI complaints and quality of life decrease.
Urogenital Distress Inventory-6 | 6 weeks
  It consists of 6 questions. In the scoring of the scale, there are options for each item: 0: not at all, 1: slightly, 2: moderately, 3: very much. Minimum 0 - maximum 18 points can be obtained from UDI-6. The score is determined by converting the points received into a percentage. An increase in the score obtained from the scale indicates that the level of quality of life is deteriorating.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Baskurt, Prof, Study Director — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data to be generated and/or analyzed during the current study are not publicly available due to confidentiality and ethical concerns, but are available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Rocha F, Carvalho J, Jorge Natal R, Viana R. Evaluation of the pelvic floor muscles training in older women with urinary incontinence: a systematic review. Porto Biomed J. 2018 Jul 18;3(2):e9. doi: 10.1016/j.pbj.0000000000000009. eCollection 2018 Oct. PMID 31595241
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Result] Bo K, Nygaard IE. Is Physical Activity Good or Bad for the Female Pelvic Floor? A Narrative Review. Sports Med. 2020 Mar;50(3):471-484. doi: 10.1007/s40279-019-01243-1. PMID 31820378
- [Result] Ghaderi F, Kharaji G, Hajebrahimi S, Pashazadeh F, Berghmans B, Pourmehr HS. Physiotherapy in Patients with Stress Urinary Incontinence: A Systematic Review and Meta-analysis. Urol Res Pract. 2023 Sep;49(5):293-306. doi: 10.5152/tud.2023.23018. PMID 37877877
- [Result] Krhut J, Zachoval R, Smith PP, Rosier PF, Valansky L, Martan A, Zvara P. Pad weight testing in the evaluation of urinary incontinence. Neurourol Urodyn. 2014 Jun;33(5):507-10. doi: 10.1002/nau.22436. Epub 2013 Jun 24. PMID 23797972
- [Result] Shin DC, Shin SH, Lee MM, Lee KJ, Song CH. Pelvic floor muscle training for urinary incontinence in female stroke patients: a randomized, controlled and blinded trial. Clin Rehabil. 2016 Mar;30(3):259-67. doi: 10.1177/0269215515578695. Epub 2015 Apr 10. PMID 25862769
- [Result] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117
- [Result] Yesil H, Akkoc Y, Karapolat H, Guler A, Sungur U, Evyapan D, Gokcay F. Reliability and validity of the Turkish version of the Danish Prostatic Symptom Score to assess lower urinary tract symptoms in stroke patients. NeuroRehabilitation. 2017;41(2):429-435. doi: 10.3233/NRE-162136. PMID 28946578
- [Result] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Result] Farzinmehr A, Moezy A, Koohpayehzadeh J, Kashanian M. A Comparative Study of Whole Body Vibration Training and Pelvic Floor Muscle Training on Women's Stress Urinary Incontinence: Three- Month Follow- Up. J Family Reprod Health. 2015 Nov;9(4):147-54. PMID 27047560
- [Result] Kannan P, Hsu WH, Suen WT, Chan LM, Assor A, Ho CM. Yoga and Pilates compared to pelvic floor muscle training for urinary incontinence in elderly women: A randomised controlled pilot trial. Complement Ther Clin Pract. 2022 Feb;46:101502. doi: 10.1016/j.ctcp.2021.101502. Epub 2021 Oct 26. PMID 34763295
- [Result] Lopes-Souza P, Dionello CF, Bernardes-Oliveira CL, Moreira-Marconi E, Marchon RM, Teixeira-Silva Y, Paineiras-Domingos LL, da Cunha Sa-Caputo D, Xavier VL, Bergmann A, Klumb EM, Bernardo-Filho M. Effects of 12-week whole-body vibration exercise on fatigue, functional ability and quality of life in women with systemic lupus erythematosus: A randomized controlled trial. J Bodyw Mov Ther. 2021 Jul;27:191-199. doi: 10.1016/j.jbmt.2021.01.015. Epub 2021 Jan 27. PMID 34391233